CLINICAL TRIAL: NCT03236857
Title: A Phase 1 Study of the Safety and Pharmacokinetics of Venetoclax in Pediatric and Young Adult Patients With Relapsed or Refractory Malignancies
Brief Title: A Study of the Safety and Pharmacokinetics of Venetoclax in Pediatric and Young Adult Patients With Relapsed or Refractory Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Collaborators: Roche-Genentech (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M13-833; 2017-000439-14 (EudraCT Number)
Expanded Access: NCT03123029 (Available)
Record Dates: First submitted 2017-07-31; First posted 2017-08-02 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2022-11

CONDITIONS: Malignancies; Acute Lymphoblastic Leukemia (ALL); Acute Myeloid Leukemia (AML); Non-Hodgkin's Lymphoma; Neuroblastoma
Keywords: Cancer; Venetoclax; pediatric; relapsed or refractory; Venclexta
MeSH Terms: conditions — Neoplasms; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Lymphoma, Non-Hodgkin; Neuroblastoma; Recurrence | interventions — Drug Therapy; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Venetoclax with or without chemotherapy (Experimental): Venetoclax administered orally once daily (QD) with various doses and dosing regimens with or without chemotherapy at the discretion of the investigator. Allowed chemotherapy regimens as outlined in the study protocol.
  Interventions: Drug: chemotherapy; Drug: venetoclax

INTERVENTIONS:
Drug: chemotherapy — Dexamethasone and/or vincristine and/or pegasparaginase OR cytarabine and/or etoposide and/or pegasparaginase; tyrosine kinase inhibitor; cytarabine OR azacitidine OR decitabine; rituximab and/or dexamethasone and/or vincristine; cyclophosphamide and/or topotecan
Drug: venetoclax — Oral tablet for participants; Tablet for oral suspension (participants who cannot swallow a tablet)
  Other Names: ABT-199; GDC-0199; Venclexta

SUMMARY:
An open-label, global, multi-center study to evaluate the safety and pharmacokinetics of venetoclax monotherapy, to determine the dose limiting toxicity (DLT) and the recommended Phase 2 dose (RPTD), and to assess the preliminary efficacy of venetoclax in pediatric and young adult participants with relapsed or refractory malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have relapsed or refractory cancer.
* Participants must have adequate hepatic and kidney function.
* Participants less than or equal to 16 years of age must have performance status of Lansky greater than or equal to 50% and participants greater than 16 years of age must have performance status of Karnofsky greater than or equal to 50%.
* Participants with solid tumors (with the exception of neuroblastoma) must have adequate bone marrow function in Part 1.
* For the fifth cohort during Part 2 Cohort Expansion, participants with solid tumors must have evidence of BCL-2 expression (except participants with TCF3-HLF ALL).

Exclusion Criteria:

* Participants with primary brain tumors or disease metastatic to the brain.
* Participants who have central nervous system (CNS) disease with cranial involvement that requires radiation.
* Participants who have received any of the following within the listed time frame, prior to the first dose of study drug

  * Inotuzumab ozogamicin or gemtuzumab ozogamicin within 30 days
  * Biologic agent (i.e., antibodies) for anti-neoplastic intent within 30 days or 5 half-lives whichever is shorter.
  * CAR-T infusion or other cellular therapy within 30 days
  * Anticancer therapy including chemotherapy, radiation therapy, targeted small molecule agents, investigational agents within 14 days or 5 half-lives, whichever is shorter (Exceptions: Ph+ALL participants on Tyrosine Kinase Inhibitor (TKI) at Screening may enroll and remain on TKI therapy to control disease and TCF3-HLF ALL participants are allowed to have received chemotherapy within 14 days or 5 half-lives, whichever is shorter).
  * Steroid therapy for anti-neoplastic intent within 5 days (with the exception of TCF3-HLF ALL participants).
  * Requires ongoing hydroxyurea (hydroxyurea permitted up to first dose)
* Participants who are less than 100 days post-transplant, or greater than or equal to 100 days post-transplant with active graft versus host disease (GVHD), or are receiving immunosuppressant therapy within 7 days prior to first dose of study drug.
* Participants who are less than 6 weeks post-131 I-metaiodobenzylguanidine (mIBG) therapy.
* Participants who have received the following within 7 days prior to the first dose of study drug:

  * Strong and moderate Cytochrome P450 3A (CYP3A) inhibitors (Part 1 Dose Determination);
  * Strong and moderate CYP3A inducers (Part 1 Dose Determination and Part 2 Cohort Expansion).
* Participants who have not recovered from clinically significant adverse effect(s)/toxicity(s) of the previous therapy (Exception: Chemotherapy induced side effects that are expected to return to baseline in TCF3-HLF ALL participants).
* Participants who have active, uncontrolled infections.
* Participants with malabsorption syndrome or any other condition that precludes enteral administration.

  * Participants with recent positive test for SARS-CoV-2 (COVID-19) and no follow up test with negative result cannot be enrolled. Participants with contact to persons with COVID-19 and participants with signs and symptoms for COVID-19 infection must be tested before enrolling.

Ages: 0 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 143 (Actual)
Dates: Start 2017-11-08 (Actual); Primary Completion 2023-04-19 (Actual); Study Completion 2023-04-19 (Actual)

PRIMARY OUTCOMES:
Number of Participants Experiencing Adverse Events | Up to 9 months
  An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment. The investigator assesses the relationship of each event to the use of study.
Number of Participants With Dose Limiting Toxicities (DLT) of Venetoclax Monotherapy | First 21 days venetoclax monotherapy
  A DLT is any Grade 3 or higher non-hematologic adverse event (AE) with exceptions outlined in the protocol.
Recommended Phase 2 dose (RPTD) of Venetoclax | First 21 days venetoclax monotherapy
  Venetoclax RPTD is the dose determined based on adverse event reporting and dose-limiting toxicity information from all participants.
Cmax of Venetoclax | Up to approximately 2 weeks
  Maximum plasma concentration (Cmax) of venetoclax.
Tmax of venetoclax | Up to approximately 2 weeks
  Time to maximum plasma concentration (Tmax) of venetoclax.
AUC0-24 Post-Dose of Venetoclax | Up to approximately 2 weeks
  Area under the plasma concentration-time curve from 0 to 24 hours (AUC24) post-dose of venetoclax.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to 9 months
  ORR is defined as the proportion of participants who achieved a response according to established criteria described in detail in the study protocol.
Partial Response (PR) Rate | Up to 9 months
  PR is defined according to established criteria for each tumor type and is described in detail within the study protocol.
Complete Response (CR) Rate | Up to 9 months
  CR is defined according to established criteria for each tumor type and is described in detail within the study protocol.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (31):
- United States (11):
  - Univ California, San Francisco /ID# 163460, San Francisco, California
  - Children's Hospital Colorado /ID# 161551, Aurora, Colorado
  - Children's Healthcare of Atlan /ID# 161552, Atlanta, Georgia
  - Dana-Farber Cancer Institute /ID# 163440, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center-Koch Center /ID# 163444, New York, New York
  - Cincinnati Children's Hospital /ID# 161550, Cincinnati, Ohio
  - Children's Hospital of Philadelphia /ID# 163445, Philadelphia, Pennsylvania
  - St Jude Children's Research Hospital /ID# 163447, Memphis, Tennessee
  - Primary Children's /ID# 164399, Salt Lake City, Utah
  - Seattle Children's Hospital /ID# 163459, Seattle, Washington
  - Medical College of Wisconsin /ID# 163461, Milwaukee, Wisconsin
- Australia (4):
  - Sydney Children's Hospital /ID# 163148, Randwick, New South Wales
  - Queensland Children's Hospital /ID# 163146, South Brisbane, Queensland
  - Women and Childrens Hospital /ID# 163147, North Adelaide, South Australia
  - Royal Children's Hospital /ID# 163104, Parkville, Victoria
- Canada (2):
  - Hospital for Sick Children /ID# 163726, Toronto, Ontario
  - CHU Sainte-Justine /ID# 163725, Montreal, Quebec
- France (5):
  - AP-HM - Hopital de la Timone /ID# 161465, Marseille, Bouches-du-Rhone
  - Centre Leon Berard /ID# 163707, Lyon, Rhone
  - AP-HP - Hopital Armand-Trousseau /ID# 163728, Paris
  - Robert Debre Hopital, FR /ID# 161464, Paris
  - CHU Toulouse - Hôpital des enfants /ID# 163727, Toulouse
- Germany (4):
  - Universitaetsklinikum Freiburg /ID# 164206, Freiburg im Breisgau, Baden-Wurttemberg
  - Universitaetsklinikum Schleswig-Holstein Campus Kiel /ID# 161729, Kiel, Schleswig-Holstein
  - Charite Universitaetsklinikum Berlin - Campus Virchow /ID# 161730, Berlin
  - Universitaetsklinikum Essen /ID# 164207, Essen
- Netherlands (2):
  - Erasmus MC - Sophia /ID# 161579, Rotterdam
  - Prinses Maxima Centrum /ID# 162670, Utrecht
- Kinderspital Zurich - Eleonorenstiftung /ID# 163037, Zurich, Canton of Zurich, Switzerland
- United Kingdom (2):
  - Great Ormond Street Hospital for Children /ID# 169238, London, London, City of
  - The Newcastle Upon Tyne Hospitals NHS Foundation Trust /ID# 162938, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Karol SE, Khaw SL, Zwaan CM, Baruchel A, Bittencourt H, Cooper TM, Flotho C, Fraser C, Forlenza CJ, Goldsmith KC, Macy ME, Morgenstern DA, O'Brien MM, Petit A, Ziegler DS, Reinhardt D, Opferman JT, Rubnitz JE, Onishi M, Dunshee DR, Dunbar F, Vishwamitra D, Ross JA, Chen X, Unnebrink K, Kammerlander M, Salem AH, Palenski TL, Sunkersett G, Place AE. Venetoclax Alone or in Combination With Chemotherapy in Paediatric and Adolescent/Young Adult Patients With Relapsed/Refractory Acute Myeloid Leukaemia. Pediatr Blood Cancer. 2025 Jul;72(7):e31714. doi: 10.1002/pbc.31714. Epub 2025 Apr 23. PMID 40266036
- [Derived] Place AE, Karol SE, Forlenza CJ, Cooper TM, Fraser C, Cario G, O'Brien MM, Gerber NU, Bourquin JP, Reinhardt D, Rubnitz JE, Opferman JT, Sunkersett G, Onishi M, Dunshee DR, Chen X, Unnebrink K, Vishwamitra D, Dunbar F, Badawi M, Ross JA, Loh ML. Venetoclax Combined With Chemotherapy in Pediatric and Adolescent/Young Adult Patients With Relapsed/Refractory Acute Lymphoblastic Leukemia. Pediatr Blood Cancer. 2025 Jun;72(6):e31630. doi: 10.1002/pbc.31630. Epub 2025 Mar 10. PMID 40062648
- [Derived] Badawi M, Gopalakrishnan S, Engelhardt B, Palenski T, Karol SE, Rubnitz JE, Menon R, Salem AH. Dosing of Venetoclax in Pediatric Patients with Relapsed Acute Myeloid Leukemia: Analysis of Developmental Pharmacokinetics and Exposure-Response Relationships. Clin Ther. 2024 Oct;46(10):759-767. doi: 10.1016/j.clinthera.2024.09.008. Epub 2024 Oct 5. PMID 39368878
- [Derived] Dalton KM, Krytska K, Lochmann TL, Sano R, Casey C, D'Aulerio A, Khan QA, Crowther GS, Coon C, Cai J, Jacob S, Kurupi R, Hu B, Dozmorov M, Greninger P, Souers AJ, Benes CH, Mosse YP, Faber AC. Venetoclax-based Rational Combinations are Effective in Models of MYCN-amplified Neuroblastoma. Mol Cancer Ther. 2021 Aug;20(8):1400-1411. doi: 10.1158/1535-7163.MCT-20-0710. Epub 2021 Jun 4. PMID 34088831
- [Derived] Place AE, Goldsmith K, Bourquin JP, Loh ML, Gore L, Morgenstern DA, Sanzgiri Y, Hoffman D, Zhou Y, Ross JA, Prine B, Shebley M, McNamee M, Farazi T, Kim SY, Verdugo M, Lash-Fleming L, Zwaan CM, Vormoor J. Accelerating drug development in pediatric cancer: a novel Phase I study design of venetoclax in relapsed/refractory malignancies. Future Oncol. 2018 Sep;14(21):2115-2129. doi: 10.2217/fon-2018-0121. Epub 2018 Mar 29. PMID 29595064